CLINICAL TRIAL: NCT03682029
Title: Epigenetics, Vitamin C, and Abnormal Hematopoiesis - Role of Vitamin C in Epigenetic Regulation in Hematopoiesis Sub-Study on CCUS, Low-Risk MDS, and CMML-0/1
Brief Title: Epigenetics, Vitamin C, and Abnormal Blood Cell Formation - Vitamin C in Patients With Low-Risk Myeloid Malignancies
Acronym: EVITA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Van Andel Institute - Stand Up To Cancer Epigenetics Dream Team (Unknown); University of Southern California (Other); Imperial College London (Other); University of Copenhagen (Other); Odense University Hospital (Other); Technical University of Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Grønbæk, Professor, MD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-16022249 low-risk cohort
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia-1; Cytopenia
Keywords: Clonal Cytopenia of Undetermined Significance; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Low-Risk Myeloid Malignancies; Vitamin C; Epigenetics; TET2; Randomized, Placebo-Controlled Trial; Clinical Study
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia; Leukemia, Myelomonocytic, Chronic | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization performed by the independent provider of study medication (Glostrup Pharmacy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Vitamin C (ascorbic acid) 500 mg/capsule. Ingestion of 2 capsules (1000 mg) daily for 12 months.
  Interventions: Dietary Supplement: Vitamin C (ascorbic acid)
- Placebo (Placebo Comparator): Placebo capsule. Ingestion of 2 capsules daily for 12 months. Placebo will be prepared as capsules that look and taste identical to the vitamin C supplement capsules. The content of the placebo is lactose, potato starch, gelatin, magnesium stearate, and talc.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C (ascorbic acid) — Monotherapy with oral vitamin C supplementation to elevate plasma vitamin C level to the upper end of the physiological range.
  Arms: Vitamin C
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this multi-centre, randomized, placebo-controlled, double-blind phase II study is to investigate if oral vitamin C may change the biology of low-risk myeloid malignancies; i.e., clonal cytopenia of undetermined significance (CCUS), low-risk myelodysplastic syndromes (MDS), and chronic myelomonocytic leukemia (CMML)-0/1 by reversing the epigenetic changes characteristic of these disease entities. The epigenetic regulator TET2 is the gene most often affected in CCUS. Preclinical studies have shown that active demethylation by the TET enzymes is dependent on vitamin C, and the investigators and collaborators have shown that plasma vitamin C levels are exceedingly low in hematological cancer patients but are easily corrected by oral vitamin C. This study is part of an array of EVITA studies aimed at clarifying whether the standard of care of patients with myeloid malignancies should be changed and oral vitamin C supplement added to the treatment recommendations.

DETAILED DESCRIPTION:
BACKGROUND Recent investigations have shown that mutations in epigenetic regulators are common, both in the apparently normal hematopoiesis of the elderly and in patients (pts) with myeloid cancers. It was long anticipated that DNA methylation was a permanent silencing mark, but with the discovery of the ten eleven translocation (TET) enzymes it became clear that active demethylation occurs. The initial steps in this process are catalyzed by TET enzymes, which are, however, frequently mutated and methylated in hematological cancers. The Jumonji enzymes, which catalyze histone demethylation, are also aberrantly regulated in hematological cancers.

Vitamin C (VitC) was identified in the 1930'ies as the necessary micronutrient in the prevention of scurvy. Unlike plants and most animals, humans are unable to synthesize vitC from glucose due to lack of the required enzyme, L-gulonolactone oxidase. Therefore, vitC must be provided through the diet. Recent studies recognize vitC as an important cofactor for the Fe(II)- and 2-oxoglutarate dioxygenase family. These include the TET enzymes, which are involved in the conversion of 5-methylcytosine (5-mC) to its oxidized derivatives 5-hydroxymethylcytosine (5-hmC), 5-carboxyl cytosine (5-caC), and 5-formylcytosine (5-fC), and the Jumonji enzymes that are involved in histone demethylation. Accordingly, vitC may potentially play an important role in the regulation of DNA and histone demethylation. However, > 80 percentage of hematological cancer pts were found to be severely vitC deficient. Interestingly, analyses of 20 participants included in the investigators' recently conducted randomized, placebo-controlled pilot study (NCT02877277) show that the level of vitC in MDS and CMML pts undergoing treatment with azacitidine, is easily elevated to the normal range by oral vitC supplement (unpublished data). When pts that were already taking vitC supplements were switched to placebo, the vitC levels quickly dropped below the normal range.

It has also been shown that the formation of 5-hmC and its derivatives may be compromised in healthy individuals and pts with TET mutations. However, since many of these mutations are heterozygous, and since the three TET enzymes (TET1, TET2, and TET3) may have some redundancy, restoration of vitC to physiological levels might have an impact on the level of 5-hmC/5-mC in individuals with TET mutant clonal hematopoiesis or hematological cancer.

Analyses of 5-hmC/5-mC levels in peripheral blood (PB) mononuclear cells (MNCs) from the participants in the pilot study also showed a clear trend toward increased 5-hmC in the vitC arm, however, after designing the trial the investigators realized that 5-hmC/5-mC levels are better measured in hematopoietic stem cells in the bone marrow (BM) where the levels are 10-20 fold higher. Thus, the pilot study will be followed-up with a randomized placebo-controlled trial of oral vitC in individuals with low-risk myeloid malignancies; i.e., CCUS or low-risk MDS/CMML, to investigate if oral vitC can change the biology of these disease entities and ultimately prevent progression.

Hypotheses:

1. The investigators and collaborators have previously shown that cancer pts are vitC deficient, and individuals with CCUS, which represents pre-MDS, might also be vitC deficient. The hypothesis is that this may lead to reduced levels of 5-hmC/5-mC in vivo in both cancer pts and individuals with CCUS
2. Elevating serum vitC levels to the normal range in CCUS and low-risk MDS/CMML pts by oral supplementation with vitC may

   * reduce the malignant clone,
   * increase the 5-hmC/5-mC ratio,
   * change the plasma cytokine profile towards a less inflammatory, less tumorigenic profile,
   * change gene expression

Aims:

To determine if restoring vitC to the normal range in CCUS and low-risk MDS/CMML pts can:

1. reduce the malignant clone,
2. increase the 5-hmC/5-mC ratio in CCUS and low-risk MDS/CMML pts
3. reduce accumulation of 5-mC at promoters/enhancers/long terminal repeats (LTRs), or at other regulatory genomic regions of tumor suppressors/methylated driver genes/genes involved in hematopoietic development,
4. upregulate the expression of these genes,
5. change the plasma cytokine profile,
6. alter intestinal permeability (measured by concentration of bacterial DNA in peripheral blood) and/or composition of gut microbiota,
7. entail any safety risks.

RESEARCH PLAN A total of 100 patients is planned for enrolment. Individuals with CCUS, low-risk MDS, or CMML-0 or -1 will be included from Rigshospitalet, Herlev University Hospital, Odense University Hospital, Aalborg University Hospital or Keck Hospital of University of Southern California between November 2017-December 2021.

The participants will enter block randomization with a ratio of 1:1; vitC 1000 mg/day p.o. versus placebo for one year.

Up to 30 healthy elderly volunteers are planned for enrolment. Amount and type of bacterial DNA in PB will be determined and serve as controls.

MATERIAL AND MEASUREMENTS PB: PB samples (45 mL) will be taken at study entry and every 3 months (or more if required according to physician's choice) during the first year.

Measurements include blood counts including differential count, levels of folic acid, vitamin B12, vitamin D, iron, ferritin, transferrin, transferrin saturation, plasma vitC levels, cytokines, and bacterial DNA content (referenced to bacterial DNA on patient's skin and in feces).

BM: BM samples (18 mL) will be taken at study entry, after 3 months, and after one year.

Levels of vitC and various cytokines will be measured. Mutations in genes frequently involved in myeloid cancer/clonal hematopoiesis, including epigenetic regulators, and variant allele frequencies (VAF) will be investigated by targeted next generation sequencing in sorted BM CD34+ cells (if available) or BM negative fraction of CD34+ sorting at study entry, after 3 months and after one year.

RNA sequencing and total 5-hmC/5-mC assessment will be performed on BM CD34+ hematopoietic stem cells.

Feces: Feces samples (9 mL) will be collected from a subset of patients at study entry, after 3 months, and after one year. Bacterial DNA will be extracted and sequenced.

RESEARCH BIOBANK A research biobank will be established at The Epi-/Genome Laboratory, Rigshospitalet / Biotech Research and Innovation Centre to store the biological samples from the participants. The research biobank is approved by the Regional Science Ethics Committee and the Danish Data Protection Agency in accordance with the Act on Processing of Personal Data (license no. H-16022249 and 04864/RH-2016-259, respectively). Cryopreserved separated MNCs from BM and PB will be stored in addition to granulocyte pellets and plasma. The date for closing the research biobank is 31-12-2030.

For correlative studies, biological samples will be sent to Van Andel Research Institute, Grand Rapids, US, and Imperial College, London, UK (external collaborators), for RNA sequencing and analyses of DNA methylation and hydroxymethylation, respectively. Biological samples will also be sent to Life Science Faculty, University of Copenhagen, and The National Veterinary Institute, Technical University of Denmark (external collaborators) for measurement of serum vitC concentrations and analyses of T cell responses, respectively.

METHODS VitC measurement: Ascorbate and total vitC, i.e., ascorbate + dehydroascorbic acid (the oxidized form of vitC; DHA), are quantified by high-performance liquid chromatography (HPLC) with coulometric detection; DHA is assessed by subtraction of ascorbate from total vitC. Uric acid is used as endogenous internal standard.

Cell sorting: Magnetic-activated cell sorting (MACS, using a EasySep device).

Total 5-hmC/5-mC measurement: Dot blot analysis of 5-hmC. 5-hmC/5-mC measurement by Mass Spectrometry.

Locus specific 5-hmC/5-mC measurement: "EPIC" 850 K BeadChips. 5-hmC/5-mC at selected sites will be measured by pyrosequencing.

Gene expression: Total RNA sequencing and reverse transcriptase-quantitative polymerase chain reaction.

Mutation detection: Targeted next generation sequencing of a panel of genes recurrently mutated in myeloid cancer as described.

STATISTICAL CONSIDERATIONS AND POWER CALCULATION This study is the first study to examine the effects of vitC as monotherapy on 5-hmC/5-mC levels in hematopoietic stem cells in humans in vivo. Therefore, it is not possible to perform a power calculation or a sample size calculation. The number of participants (n=100) is set as an estimate of the number needed to observe a potential significant difference between the groups (vitC vs. placebo) in the primary endpoint; median change in VAF of somatic mutations from baseline to 12 months.

Efficacy analyses are by intention-to-treat. Safety analyses include all participants who receive at least one dose of protocol therapy.

ETHICAL CONSIDERATIONS The study has been approved by the Regional Science Ethics Committee (H-16022249) and the Danish Data Protection Agency (04864/RH-2016-259).

All participants included in the project will be informed orally and in writing. Participation will only be accepted after written consent. Participants will be informed that they can at any time for any reason withdraw from the study without it affecting their treatment in the health care system.

Using the targeted DNA sequencing approach described, there is a small risk of detecting a germline mutation in the participants related to myeloid malignancy. The participants will be asked to state in the informed consent if they do not want to receive any further relevant health-related information that may appear during the project analyses. Unless the participant explicitly states that he or she does not want to be informed of any potential health-related random findings in the study, the participant will be informed and offered further investigations and genetic counseling at the local hospital in case of random findings.

Patient disadvantages, side effects, risks, and complications Blood sampling is associated with brief discomfort and/or pain. No significant risks are associated with the blood sampling. Local bleeding can occur, which in rare cases can cause discomfort and discoloration for a few days. Rarely, a blood sampling can cause vasovagal reaction leading to a brief loss of consciousness.

BM aspiration is associated with brief pain while the local anesthesia is given. Furthermore, many individuals experience an uncomfortable feeling in the nates and leg while the BM is aspirated. This lasts approximately 30 seconds. Finally, some tenderness can occur for a few days after the procedure. Possible complications to undergoing a BM investigation include bleeding and infection. However, the incidence of these complications is extremely low.

According to the Nordic Nutrition Recommendations there is no evidence that intake of vitC above 1000 mg/day are either carcinogenic or teratogenic. However, high intakes (> 1000-2000 mg/day) may cause diarrhea and other gastrointestinal disturbances and susceptible individuals may experience kidney stone formation from increased oxalate formation. Since vitC is only given at physiological doses, it is anticipated that the study is safe and will provide no additional risk for the participants; an assumption that is supported by the experience from the pilot study.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of CCUS:

* Persistent cytopenia for > 6 months defined as hgb < 11.3 g/dL (7 mmol/L) in women and hgb < 12.9 g/dL (8 mmol/L) in men, thrombocyte count < 150 x 10^9/L or neutrophil count < 1.8 x 10^9/L
* Normal cytogenetics (with the exception of deletion of the Y chromosome which can be accepted)
* A bone marrow morphology that is not diagnostic of MDS or any other malignancy
* Other common causes of cytopenia (vitamin or other deficiencies, virus infection, etc.) have been ruled out
* Hematolytic conditions have been ruled out
* The presence of a detectable mutation in genes recurrently affected in myeloid malignancy representing a clonal marker (excluding germline mutations)

OR

A diagnosis of MDS as according to World Health Organization (WHO) 2016 diagnostic criteria

• Revised international prognostic scoring system (IPSS-R) risk score ≤ 3 AND bone marrow blast percentage < 5 defining low-risk

OR

A diagnosis of CMML-0 or -1 as according to WHO 2016 diagnostic criteria

AND

(All diagnostic categories) The presence of a detectable mutation in genes recurrently affected in myeloid malignancy representing a clonal marker (excluding germline mutations)

Exclusion Criteria:

* Unwillingness to discontinue any and all use of vitamin C medication/supplementation including multivitamin at least 24 hours prior to Baseline investigations and sampling
* Lack of ability to understand the information given, or lack of willingness to sign a written informed consent document
* Treatment with chemotherapy within the past 6 months
* Patients receiving active treatment for their myeloid malignancy, including investigational agents, with the exception of granulocyte colony-stimulating factor (G-CSF) and erythropoietin
* History of allergic reactions to ascorbic acid
* Unwillingness to comply with all aspects of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2025-09-27 (Estimated)

PRIMARY OUTCOMES:
Median Change from Baseline in Variant Allele Frequency at 12 Months | At baseline and at 12 months
  Median change from baseline to 12 months in mutant allele burden as measured by the variant allele frequency (VAF) and number of mutations in the vitC group vs. the placebo group.

SECONDARY OUTCOMES:
Mean Change from Baseline in 5-hmC/5-mC Level at 3 Months and 12 months | At baseline and at 3 months and 12 months
  Mean change from baseline to 3 months and 12 months in global 5-hmC/5-mC measured in hematopoietic stem cells is compared between the vitamin C group and the placebo group. In addition, the mean change from baseline in 5-hmC/5-mC at 12 months is compared between participants in the vitamin C arm with baseline plasma vitamin C level in the normal range vs. participants in the vitamin C arm with baseline plasma vitamin C level below the normal range.
Mean Change from Baseline in 5-mC at Selected Sites at 12 Months | At baseline and at 12 months
  Mean change from baseline to 12 months in 5-mC at promoters/enhancers/long terminal repeats, and other regulatory genomic regions of tumor suppressors/methylated driver genes/genes involved in hematopoietic development.
Mean Change from Baseline in H3K9 Methylation at Selected Sites at 12 Months | At baseline and at 12 months
  Mean change from baseline to 12 months in methylated histone H3 lysine at position 9 at promoters/enhancers/long terminal repeats, and other regulatory regions of tumor suppressors/methylated driver genes/genes involved in hematopoietic development.
Mean Change from Baseline in Plasma Cytokine Levels at 12 Months | At baseline and at 12 months
  Mean change from baseline to 12 months in plasma cytokine levels (e.g., IL-6, S100A9, etc.).
Mean Change from Baseline in mRNA Levels of Selected Genes at 12 Months | At baseline and at 12 months
  Mean change from baseline to 12 months in mRNA levels of tumor suppressor genes, oncogenes, epigenetic regulators, cytokines, and genes involved in hematopoietic development.
Mean Change from Baseline in mRNA Levels of Selected Genes at 3 Months | At baseline and at 3 months
  Mean change from baseline to 3 months in mRNA levels of tumor suppressor genes, oncogenes, epigenetic regulators, cytokines, and genes involved in hematopoietic development.
Number of Participants with Serious Adverse Events and Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Through study completion, 12 months
  Number of serious adverse events and treatment-related adverse events as assessed by CTCAE v5.0. Adverse events, that are not considered serious or related to vitamin C intake, will not be recorded.
Percentage of Participants with Vitamin C Deficiency | Day 1
  Percentage of participants with baseline plasma vitamin C level below the normal physiological range.
Change in intestinal permeability and gut microbiota | At baseline and at 3 months and 12 months
  Change in intestinal permeability and gut microbiota (concentration of bacterial DNA in PB and adscription of bacteria by sequencing)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Grønbæk, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (5):
- Keck Hospital of University of Southern California, Los Angeles, California, United States
- Denmark (4):
  - Rigshospitalet, Copenhagen, N/A = Not Applicable
  - Aalborg University Hospital, Aalborg
  - Herlev University Hospital, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busque L, Mio R, Mattioli J, Brais E, Blais N, Lalonde Y, Maragh M, Gilliland DG. Nonrandom X-inactivation patterns in normal females: lyonization ratios vary with age. Blood. 1996 Jul 1;88(1):59-65. PMID 8704202
- [Background] Genovese G, Kahler AK, Handsaker RE, Lindberg J, Rose SA, Bakhoum SF, Chambert K, Mick E, Neale BM, Fromer M, Purcell SM, Svantesson O, Landen M, Hoglund M, Lehmann S, Gabriel SB, Moran JL, Lander ES, Sullivan PF, Sklar P, Gronberg H, Hultman CM, McCarroll SA. Clonal hematopoiesis and blood-cancer risk inferred from blood DNA sequence. N Engl J Med. 2014 Dec 25;371(26):2477-87. doi: 10.1056/NEJMoa1409405. Epub 2014 Nov 26. PMID 25426838
- [Background] Jaiswal S, Fontanillas P, Flannick J, Manning A, Grauman PV, Mar BG, Lindsley RC, Mermel CH, Burtt N, Chavez A, Higgins JM, Moltchanov V, Kuo FC, Kluk MJ, Henderson B, Kinnunen L, Koistinen HA, Ladenvall C, Getz G, Correa A, Banahan BF, Gabriel S, Kathiresan S, Stringham HM, McCarthy MI, Boehnke M, Tuomilehto J, Haiman C, Groop L, Atzmon G, Wilson JG, Neuberg D, Altshuler D, Ebert BL. Age-related clonal hematopoiesis associated with adverse outcomes. N Engl J Med. 2014 Dec 25;371(26):2488-98. doi: 10.1056/NEJMoa1408617. Epub 2014 Nov 26. PMID 25426837
- [Background] Shih AH, Abdel-Wahab O, Patel JP, Levine RL. The role of mutations in epigenetic regulators in myeloid malignancies. Nat Rev Cancer. 2012 Sep;12(9):599-612. doi: 10.1038/nrc3343. Epub 2012 Aug 17. PMID 22898539
- [Background] Tahiliani M, Koh KP, Shen Y, Pastor WA, Bandukwala H, Brudno Y, Agarwal S, Iyer LM, Liu DR, Aravind L, Rao A. Conversion of 5-methylcytosine to 5-hydroxymethylcytosine in mammalian DNA by MLL partner TET1. Science. 2009 May 15;324(5929):930-5. doi: 10.1126/science.1170116. Epub 2009 Apr 16. PMID 19372391
- [Background] Pastor WA, Aravind L, Rao A. TETonic shift: biological roles of TET proteins in DNA demethylation and transcription. Nat Rev Mol Cell Biol. 2013 Jun;14(6):341-56. doi: 10.1038/nrm3589. PMID 23698584
- [Background] Cimmino L, Dawlaty MM, Ndiaye-Lobry D, Yap YS, Bakogianni S, Yu Y, Bhattacharyya S, Shaknovich R, Geng H, Lobry C, Mullenders J, King B, Trimarchi T, Aranda-Orgilles B, Liu C, Shen S, Verma AK, Jaenisch R, Aifantis I. TET1 is a tumor suppressor of hematopoietic malignancy. Nat Immunol. 2015 Jun;16(6):653-62. doi: 10.1038/ni.3148. Epub 2015 Apr 13. PMID 25867473
- [Background] Monfort A, Wutz A. Breathing-in epigenetic change with vitamin C. EMBO Rep. 2013 Apr;14(4):337-46. doi: 10.1038/embor.2013.29. Epub 2013 Mar 15. PMID 23492828
- [Background] Grzybowski A, Pietrzak K. Albert Szent-Gyorgyi (1893-1986): the scientist who discovered vitamin C. Clin Dermatol. 2013 May-Jun;31(3):327-31. doi: 10.1016/j.clindermatol.2012.08.001. PMID 23738385
- [Background] Nishikimi M, Fukuyama R, Minoshima S, Shimizu N, Yagi K. Cloning and chromosomal mapping of the human nonfunctional gene for L-gulono-gamma-lactone oxidase, the enzyme for L-ascorbic acid biosynthesis missing in man. J Biol Chem. 1994 May 6;269(18):13685-8. PMID 8175804
- [Background] Blaschke K, Ebata KT, Karimi MM, Zepeda-Martinez JA, Goyal P, Mahapatra S, Tam A, Laird DJ, Hirst M, Rao A, Lorincz MC, Ramalho-Santos M. Vitamin C induces Tet-dependent DNA demethylation and a blastocyst-like state in ES cells. Nature. 2013 Aug 8;500(7461):222-6. doi: 10.1038/nature12362. Epub 2013 Jun 30. PMID 23812591
- [Background] Liu M, Ohtani H, Zhou W, Orskov AD, Charlet J, Zhang YW, Shen H, Baylin SB, Liang G, Gronbaek K, Jones PA. Vitamin C increases viral mimicry induced by 5-aza-2'-deoxycytidine. Proc Natl Acad Sci U S A. 2016 Sep 13;113(37):10238-44. doi: 10.1073/pnas.1612262113. Epub 2016 Aug 29. PMID 27573823
- [Background] Ko M, Huang Y, Jankowska AM, Pape UJ, Tahiliani M, Bandukwala HS, An J, Lamperti ED, Koh KP, Ganetzky R, Liu XS, Aravind L, Agarwal S, Maciejewski JP, Rao A. Impaired hydroxylation of 5-methylcytosine in myeloid cancers with mutant TET2. Nature. 2010 Dec 9;468(7325):839-43. doi: 10.1038/nature09586. PMID 21057493
- [Background] Agathocleous M, Meacham CE, Burgess RJ, Piskounova E, Zhao Z, Crane GM, Cowin BL, Bruner E, Murphy MM, Chen W, Spangrude GJ, Hu Z, DeBerardinis RJ, Morrison SJ. Ascorbate regulates haematopoietic stem cell function and leukaemogenesis. Nature. 2017 Sep 28;549(7673):476-481. doi: 10.1038/nature23876. Epub 2017 Aug 21. PMID 28825709
- [Background] Lykkesfeldt J. Ascorbate and dehydroascorbic acid as reliable biomarkers of oxidative stress: analytical reproducibility and long-term stability of plasma samples subjected to acidic deproteinization. Cancer Epidemiol Biomarkers Prev. 2007 Nov;16(11):2513-6. doi: 10.1158/1055-9965.EPI-07-0639. PMID 18006947
- [Background] Hansen JW, Westman MK, Sjo LD, Saft L, Kristensen LS, Orskov AD, Treppendahl M, Andersen MK, Gronbaek K. Mutations in idiopathic cytopenia of undetermined significance assist diagnostics and correlate to dysplastic changes. Am J Hematol. 2016 Dec;91(12):1234-1238. doi: 10.1002/ajh.24554. Epub 2016 Nov 8. PMID 27717004
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453